CLINICAL TRIAL: NCT00389467
Title: Mechanical Retrieval and Recanalization of Stroke Clots Using Embolectomy
Acronym: MR RESCUE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Chelsea S. Kidwell, MD, Professor of Neurology, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P50NS044378 (NIH); NCT00389467 (Registry Identifier: ClinicalTrials.gov); NCT00094588 (obsolete NCT alias)
Record Dates: First submitted 2006-10-16; First posted 2006-10-18 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-02

CONDITIONS: Stroke
Keywords: stroke; ischemic stroke; blood clot; Merci Retriever; Penumbra System; embolectomy; magnetic resonance imaging; MRI; CT; SPOTRIAS
MeSH Terms: conditions — Stroke; Ischemic Stroke; Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Mechanical Embolectomy (Active Comparator): Participants will be randomized to receive mechanical embolectomy treatment either with the Merci Retriever or Penumbra System and standard medical care or treatment with standard medical care alone.
  Interventions: Device: Merci Retriever and Penumbra System
- 2 (No Intervention): standard medical care

INTERVENTIONS:
Device: Merci Retriever and Penumbra System — The MERCI (Mechanical Embolus Removal in Cerebral Ischemia) Retriever consists of a flexible, nickel titanium (nitinol) wire with a helical-shaped distal tip. The helical distal tip is covered with a platinum radiopaque coil, which facilitates fluoroscopic visualization. The body of the MERCI Retriever is covered with a hydrophilic coating that helps facilitate device placement. The MERCI Retriever is available in 6 configurations (Merci Retrievers X6, L5, L4, L6, V series, DAC).
  The Penumbra System uses a reperfusion catheter in parallel with a separator component and an aspiration source to achieve separation of the thrombus and subsequent aspiration of the occlusion from the vessel. The system is available in different sizes according to the target vessels (041 Reperfusion Catheter/Separator pair for use in vessels larger than 3mm, notably the ICA and M1; 032 Reperfusion Catheter/Separator pair for use in vessels 2mm - 3mm, notably the M2).
  Arms: 1 Mechanical Embolectomy

SUMMARY:
The purpose of this study is to compare the effectiveness of treating acute ischemic stroke with mechanical embolectomy using the Merci Retriever or the Penumbra System within 8 hours of symptom onset to standard medical treatment, and to identify people who might benefit from mechanical embolectomy by the appearance of stroke on multimodal computerized tomography (CT) or magnetic resonance (MR) imaging.

DETAILED DESCRIPTION:
Stroke most commonly occurs when there is a blockage of blood flow to one of the arteries in the brain. The blockage is often caused by a clot. There is currently only one FDA-approved stroke treatment. However, only 2 percent of ischemic stroke patients receive this treatment because it must be given within 4.5 hours of the stroke onset. There is an overwhelming need for new treatments that extend the time window to treatment since most individuals with stroke arrive at the hospital after the 4.5-hour time window.

Two of the most promising new devices are the Merci Retriever, a tiny corkscrew device, and the Penumbra System, an aspiration device. Both are designed to remove clots from arteries and thereby restore blood flow to the brain.

The primary purpose of this study is to compare the effectiveness of treatment with the Merci Retriever or Penumbra System within 8 hours of symptom onset to standard medical treatment, and to identify people who might benefit from the devices by the appearance of the stroke on multimodal computerized tomography (CT) or magnetic resonance imaging (MRI). Previous testing has determined that the use of the Merci Retriever is successful in opening up blocked blood vessels in approximately ½ of the individuals in whom it is used, and the Penumbra System is successful in opening up blocked blood vessels in approximately 80% of the individuals in whom it is used.

A total of 120 participants from approximately 30 different medical centers will be enrolled into this study. Participants will be randomized to either receive treatment by mechanical embolectomy with the Merci Retriever or Penumbra System and standard medical care or treatment with standard medical care alone. Standard care for stroke patients may include intravenous fluid, careful regulation of blood pressure, blood-thinning medicine (such as heparin or warfarin), anti-platelet medicine (such as aspirin or clopidogrel), and rehabilitation therapies.

Participants undergoing the Merci Retriever or Penumbra System procedure will have a cerebral arteriogram with pictures taken with dye prior to the procedure to determine the location of the blockage, and following the procedure to determine if blood supply has been restored. The total mechanical embolectomy procedure with either device will take approximately 1 to 2 hours. Participants will have brief neurological exams several times during this time to monitor changes in their neurological condition.

Participants will have follow-up visits, including neurological exams, at 30 days and at 90 days.

This study is part of the Specialized Program of Translational Research in Acute Stroke (SPOTRIAS), which allows researchers to enhance and initiate translational research that ultimately will benefit stroke patients by treating more patients in less than 2 hours, and finding ways to treat additional patients later.

ELIGIBILITY:
Inclusion Criteria:

* New focal disabling neurologic deficit consistent with acute cerebral ischemia (NIHSS >/= 6)
* Age >/= 18 ≤ 85
* Clot retrieval procedure can be initiated within 8 hours from onset
* Large vessel proximal anterior circulation occlusion on MR or CT angiography (internal carotid, M1 or M2 MCA)
* Pretreatment MRI performed according to MR RESCUE protocol
* Signed informed consent obtained from the patient or patient's legally authorized representative
* Premorbid modified Rankin score of 0-2
* Allowed but not required: patients treated with IV tPA (tissue plasminogen activator) up to 4.5 hours from symptom onset with persistent target occlusion on post-treatment MR RESCUE MR or CT protocol performed at the completion of drug infusion (Note: Rapidly improving neurological signs prior to randomization is an exclusion)

Exclusion Criteria:

* NIHSS >/= 30
* Contraindication to MRI (pacemaker etc)
* Acute intracranial hemorrhage
* Coma
* Rapidly improving neurological signs prior to randomization
* Pre-existing medical, neurological or psychiatric disease that would confound the neurological, functional, or imaging evaluations
* Pregnancy
* Known allergy to iodine previously refractory to pretreatment medications
* Current participation in another experimental treatment protocol
* Contrast-Enhanced Neck MRA (magnetic resonance angiography) or CTA (computed tomography angiography) suggests proximal ICA occlusion, proximal carotid stenosis > 67%, or dissection
* INR > 3.0 (international normalized ratio)
* PTT > 3 x Normal (partial thromboplastin time)
* Imaging data cannot be processed by the MR RESCUE computer
* Renal Failure (serum creatinine > 2.0 or Glomerular Filtration Rate [GFR] < 30)

MRI Exclusion Criteria:

* Contraindication to MRI (pacemaker, etc)

CT Exclusion Criteria:

* Contraindication to iodinated contrast**

  **Examples of possible iodinated contrast contraindications include:
* Hyperthyroidism
* History of severe allergic reaction to iodinated contrast material
* History of sever kidney disease as an adult, including tumor or transplant surgery, or family history of kidney failure
* Paraproteinemia syndromes or multiple myeloma
* Collagen vascular disease
* Severe cardiac insufficiency
* Severely compromised liver function
* Current therapy with metformin, aminoglycosides

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2004-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea S Kidwell, MD, Principal Investigator — Professor of Neurology, Georgetown University; Reza Jahan, MD, Principal Investigator — Associate Professor of Radiology, UCLA Medical Center, Interventional Neuroradiology
Locations (22):
- United States (21):
  - University of California at Los Angeles, UCLA Stroke Network, 924 Westwood Blvd #300, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center 4867 W Sunset Blvd., Los Angeles CA 90027, Los Angeles, California
  - Cedars Sinai Medical Center 8700 Beverly Blvd., Los Angeles CA 90048, Los Angeles, California
  - University of California at San Diego, UCSD Medical Center, 200 W. Arbor Drive, OPC, 3rd Floor Suite 3, San Diego, California
  - Santa Monica-UCLA Medical Center, 1225 15th Street Santa Monica, CA 90404, Santa Monica, California
  - Georgetown University, Georgetown University Hospital, Room GG012, Ground Floor Gorman, 3800 Reservoir Road, NW, Washington D.C., District of Columbia
  - Washington Hospital Center, 110 Irving Street, NW, Washington, DC 20010, Washington D.C., District of Columbia
  - University of Miami 1400 NW 10th Street, 10th Floor, Miami FL 33136, Miami, Florida
  - University of Iowa Hospitals and Clinics, 200 Hawkins Dr, Iowa City, IA 52242, Iowa City, Iowa
  - Suburban Hospital, 8600 Old Georgetown Road, Bethesda, MD 20814, Bethesda, Maryland
  - Boston University, One Boston Medical Center Place, Department of Neurology, C329, Boston, Massachusetts
  - Massachusetts General Hospital, 101 Huntington Ave Ste 300, Boston, Massachusetts
  - St. Louis University Hospital, 3635 Vista Avenue at Grand Boulevard Saint Louis, MO, St Louis, Missouri
  - Cornell University, New York Presbyterian Hospital, Cornell Campus, 525 East 68th St, Box 141, New York, New York
  - Columbia University, 710 W 168th St, NI 551, ,, New York, New York
  - University of Cincinnati, Department of Neurology, University of Cincinnati Medical Center, 231 Albert Sabin Way, Medical Sciences Bldg, Rm 4015, PO Box 670525, Cincinnati, Ohio
  - University of Pittsburgh, PUHC-426, 200 Lothrop Street, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, 171 Ashley Avenue, Charleston, SC 29403, Charleston, South Carolina
  - Chattanooga Center for Neurologic Research, Chattanooga, Tennessee
  - University of Texas at Houston, University of Texas, Houston Stroke Program, Department of Neurology, 6431 Fannin Street, MSB 7044, Houston, Texas
  - West Virginia University 1 Medical Center, Morgantown WV 26506, Morgantown, West Virginia
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Nael K, Knitter JR, Jahan R, Gornbein J, Ajani Z, Feng L, Meyer BC, Schwamm LH, Yoo AJ, Marshall RS, Meyers PM, Yavagal DR, Wintermark M, Liebeskind DS, Guzy J, Starkman S, Saver JL, Kidwell CS. Multiparametric Magnetic Resonance Imaging for Prediction of Parenchymal Hemorrhage in Acute Ischemic Stroke After Reperfusion Therapy. Stroke. 2017 Mar;48(3):664-670. doi: 10.1161/STROKEAHA.116.014343. Epub 2017 Jan 30. PMID 28138001
- [Derived] Kidwell CS, Jahan R, Gornbein J, Alger JR, Nenov V, Ajani Z, Feng L, Meyer BC, Olson S, Schwamm LH, Yoo AJ, Marshall RS, Meyers PM, Yavagal DR, Wintermark M, Guzy J, Starkman S, Saver JL; MR RESCUE Investigators. A trial of imaging selection and endovascular treatment for ischemic stroke. N Engl J Med. 2013 Mar 7;368(10):914-23. doi: 10.1056/NEJMoa1212793. Epub 2013 Feb 8. PMID 23394476

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2004 to 2011, participants were enrolled at 22 sites with expertise in acute stroke care, imaging and interventional neuroradiological procedures. Eligible patients presenting within 8 hours of symptom onset were enrolled. The study website generated a randomized treatment assignment using a penumbral pattern code based on brain imaging.
Pre-assignment Details: Randomization was stratified by favorable penumbral or non-penumbral pattern based on on-site analysis of baseline multimodal MRI or multimodal CT. While 127 subjects were enrolled, only 118 of these subjects qualified for the primary analysis per discussion with the DSMB as 9 subjects enrolled did not actually meet full eligibility criteria.
Groups:
- Embolectomy, Penumbral: Embolectomy patients were treated up to 8 hours from symptom onset with any combination of FDA-cleared embolectomy devices, including the Merci Retriever since trial initiation in 2004 and Penumbra System since 2009. A favorable penumbral pattern was defined as a predicted infarct core of 90 ml or less and a proportion of predicted infarct tissue within the at-risk region of 70% or less.
  Intra-arterial tPA up to 14 milligrams was allowed as rescue therapy within 6 hours of onset.
- Standard Care, Penumbral: Standard medical care was recommended per the AHA (American Heart Association)/ASA (American Stroke Association) Guidelines for management of acute ischemic stroke. A favorable penumbral pattern was defined as a predicted infarct core of 90 ml or less and a proportion of predicted infarct tissue within the at-risk region of 70% or less.
  Intra-arterial tPA up to 14 milligrams was allowed as rescue therapy within 6 hours of onset.
- Embolectomy, Nonpenumbral: Embolectomy patients were treated up to 8 hours from symptom onset with any combination of FDA-cleared embolectomy devices, including the Merci Retriever since trial initiation in 2004 and Penumbra System since 2009. A nonpenumbral pattern was defined as a predicted infarct core of greater than 90 ml or a proportion of predicted infarct tissue within the at-risk region of greater than 70%.
  Intra-arterial tPA up to 14 milligrams was allowed as rescue therapy within 6 hours of onset.
- Standard Care, Nonpenumbral: Standard medical care was recommended per the AHA (American Heart Association)/ASA (American Stroke Association) Guidelines for management of acute ischemic stroke. A nonpenumbral pattern was defined as a predicted infarct core of greater than 90 ml or a proportion of predicted infarct tissue within the at-risk region of greater than 70%.
  Intra-arterial tPA up to 14 milligrams was allowed as rescue therapy within 6 hours of onset.
Period: Overall Study
Arm/Group | Embolectomy, Penumbral | Standard Care, Penumbral | Embolectomy, Nonpenumbral | Standard Care, Nonpenumbral
Started | 34 | 34 | 30 | 20
Completed | 34 | 34 | 30 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Embolectomy, Penumbral: Treatment assignment = embolectomy, imaging pattern = penumbral
- Standard Care, Penumbral: Treatment assignment = standard medical care, imaging pattern = penumbral
- Embolectomy, Nonpenumbral: Treatment assignment = embolectomy, imaging pattern = nonpenumbral
- Standard Care, Nonpenumbral: Treatment assignment = standard medical care, imaging pattern = nonpenumbral
- Total: Total of all reporting groups
Arm/Group | Embolectomy, Penumbral | Standard Care, Penumbral | Embolectomy, Nonpenumbral | Standard Care, Nonpenumbral | Total
Number analyzed (Participants) | 34 | 34 | 30 | 20 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 12 | 16 | 7 | 51
  >=65 years | 18 | 22 | 14 | 13 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (13.2) | 65.8 (16.9) | 61.6 (12.0) | 69.4 (15.9) | 65.5 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 17 | 8 | 61
  Male | 17 | 15 | 13 | 12 | 57
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 30 | 19 | 117
  Canada | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Modified Rankin Scale Score
Description: Scale name is provided (Modified Rankin Scale) which is a standard measure of functional neurologic outcome in stroke. The scale runs from 0-6, running from perfect health without symptoms to death.
  * 0 - No symptoms.
  * 1 - No significant disability. Able to carry out all usual activities, despite some symptoms.
  * 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  * 3 - Moderate disability. Requires some help, but able to walk unassisted.
  * 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  * 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  * 6 - Dead.
Time Frame: at 90 days post-stroke
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Embolectomy, Penumbral: Embolectomy patients were treated up to 8 hours from symptom onset with any combination of FDA-cleared embolectomy devices, including the Merci Retriever since trial initiation in 2004 and Penumbra System since 2009. A favorable penumbral pattern was defined as a predicted infarct core of 90 ml or less and a proportion of predicted infarct tissue within the at-risk region of 70% or less.
- Standard Care, Penumbral: Standard medical care was recommended per the AHA (American Heart Association)/ASA (American Stroke Association) Guidelines for management of acute ischemic stroke. A favorable penumbral pattern was defined as a predicted infarct core of 90 ml or less and a proportion of predicted infarct tissue within the at-risk region of 70% or less.
- Embolectomy, Nonpenumbral: Embolectomy patients were treated up to 8 hours from symptom onset with any combination of FDA-cleared embolectomy devices, including the Merci Retriever since trial initiation in 2004 and Penumbra System since 2009. A nonpenumbral pattern was defined as a predicted infarct core of greater than 90 ml or a proportion of predicted infarct tissue within the at-risk region of greater than 70%.
- Standard Care, Nonpenumbral: Standard medical care was recommended per the AHA (American Heart Association)/ASA (American Stroke Association) Guidelines for management of acute ischemic stroke. A nonpenumbral pattern was defined as a predicted infarct core of greater than 90 ml or a proportion of predicted infarct tissue within the at-risk region of greater than 70%.
Arm/Group | Embolectomy, Penumbral | Standard Care, Penumbral | Embolectomy, Nonpenumbral | Standard Care, Nonpenumbral
Number analyzed (Participants) | 34 | 34 | 30 | 20
units on a scale | 3.9 [3.3 to 4.4] | 3.4 [2.8 to 4.0] | 4.0 [3.4 to 4.6] | 4.4 [3.6 to 5.2]

2. Secondary Outcome: Symptomatic Hemorrhagic Transformation
Description: Symptomatic intracranial hemorrhage is defined as 4 point neurologic worsening on the National Institutes of Health Stroke Scale (NIHSS) score associated with parenchymal hematoma type 2 (PH-2*), remote intracerebral hemorrhage, subarachnoid hemorrhage, or intraventricular hemorrhage on imaging. The NIHSS is a scale measuring specific neurologic deficits caused by a stroke with scores ranging from 0 to 42, and higher scores indicating more severe neurologic deficits.
  *from the modified European Cooperative Acute Stroke Study (ECASS) II criteria
Time Frame: from baseline to day 7
Measure: Number; unit: participants
Arm/Group | Embolectomy, Penumbral | Standard Care, Penumbral | Embolectomy, Nonpenumbral | Standard Care, Nonpenumbral
Number analyzed (Participants) | 34 | 34 | 30 | 20
participants | 3 | 2 | 0 | 0

3. Secondary Outcome: Day 90 Mortality
Time Frame: at day 90
Measure: Number; unit: participants
Arm/Group | Embolectomy, Penumbral | Standard Care, Penumbral | Embolectomy, Nonpenumbral | Standard Care, Nonpenumbral
Number analyzed (Participants) | 34 | 34 | 30 | 20
participants | 6 | 7 | 6 | 6

ADVERSE EVENTS:
Description: Other Adverse Events were not collected.
Arm/Group | Total Cohort | Embolectomy, Penumbral | Standard Care, Penumbral | Embolectomy, Nonpenumbral | Standard Care, Nonpenumbral
Serious Adverse Events (participants affected / at risk) | 74/118 | 25/34 | 15/34 | 22/30 | 12/20
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Total Cohort (N=118) | Embolectomy, Penumbral (N=34) | Standard Care, Penumbral (N=34) | Embolectomy, Nonpenumbral (N=30) | Standard Care, Nonpenumbral (N=20)
Neurological worsening or cerebral edema (Nervous system disorders) | 39 (41) | 11 (11) | 6 (6) | 15 (17) | 7 (7)
Procedural Complications (Nervous system disorders) | 7/64 (7) | 5 (5) | 0 (0) | 2 (2) | 0 (0)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 2 (2) | 0 (0) | 5 (6) | 2 (2)
Cardiac (Cardiac disorders) | 9 (11) | 4 (5) | 2 (3) | 2 (2) | 1 (1)
New Stroke (Nervous system disorders) | 6 (6) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Infectious (Infections and infestations) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Symptomatic Hemorrhage (Nervous system disorders) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Renal (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
DVT (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heparin Induced Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoas Hematoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amputation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 24 (24) | 5 (5) | 7 (7) | 6 (6) | 6 (6)
Asymptomatic Hemorrhage (Nervous system disorders) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No